CLINICAL TRIAL: NCT05032248
Title: Uses of Tacrolimus in Treatment of Oral Ulcers in Behcet Disease
Brief Title: Uses of Tacrolimus in Behcet Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, assistant, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: behcet
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Oral Ulcer; Behcet Syndrome
MeSH Terms: conditions — Oral Ulcer; Behcet Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tacrolimus (Experimental): group I (Colchicine and topically applied Tacrolimus),
  Interventions: Drug: Tacrolimus ointment
- placebo (Placebo Comparator): group II (Colchicine and topically applied Placebo),
  Interventions: Drug: Tacrolimus ointment

INTERVENTIONS:
Drug: Tacrolimus ointment — oral gel

SUMMARY:
Background: oral ulceration is the earliest and commonest manifestation of Behcet's disease (BD). Minor aphthous like ulcers (<10 mm in diameter) are the most common type (85%); major or herpetiform ulcers are less frequent. It is occurred about in Egypt; 3.6/100,000 % and high recurrence rate with traditional treatment. Colchicine is the first line of treatment in mucocutaneous manifestation of BD through its anti-inflammatory effect. Tacrolimus oral gel is safe and effective in treating aphthous ulcers in many diseases. Objectives: to compare the clinical efficacy of topical tacrolimus versus oral colchicine upon disease activity, pain and ulcer severity in oral ulcer associated with BD. Study design: A randomized double -blinded trial.

Setting: Rheumatology clinic, Assiut University Hospital and Faculty of Dental Medicine, AlAzhar University, Assiut branch outpatient's clinic. Methods: 40 BD participants (> 3 months taken traditional treatment with persistent active oral ulceration). They have been equally randomized into either group I (Colchicine and topically applied Tacrolimus), or group II (Colchicine only). Measurements: Behcet's Disease Current Activity Form (BDCAF), Ulcer Severity Score (USS) and visual analog scale (VAS) pre-injection, then re-evaluated postinjection at four-time points (15 days, 1st, 2nd and 3rd months) and Determination of Natural Killer (NK) cells number in salival wash before treatment (at base line) and after the treatment (after 3 months)

DETAILED DESCRIPTION:
Background: oral ulceration is the earliest and commonest manifestation of Behcet's disease (BD). Minor aphthous like ulcers (<10 mm in diameter) are the most common type (85%); major or herpetiform ulcers are less frequent. It is occurred about in Egypt; 3.6/100,000 % and high recurrence rate with traditional treatment. Colchicine is the first line of treatment in mucocutaneous manifestation of BD through its anti-inflammatory effect. Tacrolimus oral gel is safe and effective in treating aphthous ulcers in many diseases. Objectives: to compare the clinical efficacy of topical tacrolimus versus oral colchicine upon disease activity, pain and ulcer severity in oral ulcer associated with BD. Study design: A randomized double -blinded trial.

Setting: Rheumatology clinic, Assiut University Hospital and Faculty of Dental Medicine, AlAzhar University, Assiut branch outpatient's clinic. Methods: 40 BD participants (> 3 months taken traditional treatment with persistent active oral ulceration). They have been equally randomized into either group I (Colchicine and topically applied Tacrolimus), or group II (Colchicine only). Measurements: Behcet's Disease Current Activity Form (BDCAF), Ulcer Severity Score (USS) and visual analog scale (VAS) pre-injection, then re-evaluated postinjection at four-time points (15 days, 1st, 2nd and 3rd months) and Determination of Natural Killer (NK) cells number in salival wash before treatment (at base line) and after the treatment (after 3 months)

ELIGIBILITY:
Inclusion Criteria:

* active oral ulcers for Behcet's Disease

Exclusion Criteria:

* patients who received biological therapy comorbid systemic diseases allergy to Tarcolimus drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Ulcer Severity Score (USS) | 3 months
  Ulcer Severity Score (USS)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt